CLINICAL TRIAL: NCT05424939
Title: Management of Obstructive Colon Tumors in Istanbul: Multicenter Prospective Observational Cohort
Brief Title: Management of Obstructive Colon Tumors in Istanbul
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E-10840098-772.02-1214
Record Dates: First submitted 2022-05-11; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Colon Cancer; Tumor Obstruction; Emergencies; Quality of Life
MeSH Terms: conditions — Colonic Neoplasms; Emergencies | interventions — Colectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Colectomy — Colon resection
Procedure: Stoma procedures — Any type of colostomy or ileostomy with or without bowel resection
Procedure: By-pass/laparotomy/laparoscopy/biopsy — Any palliative surgery without bowel resection

SUMMARY:
The aim of this study is to evaluate the outcome of obstructive colon cancer surgery in terms of days-to-starting adjuvant therapy and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Acute intestinal obstruction due to colon cancer either preoperatively or intraoperatively detected
* Clinical findings of obstruction (Abdominal distention and pain, nausea or vomiting, and absence of bowel movements) confirmed by abdominal x-ray or CT

Exclusion Criteria:

* Benign diseases
* Emergency surgery due to bleeding, perforation and other non-obstructive situations
* Recurrent colon tumors
* Rectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who underwent surgery with a clinical and radiological diagnosis of obstructive colon tumors at any stage will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Time-to-starting chemotherapy | 1 year
  Surgical procedures will be compared in terms of days-to-first chemotherapy

SECONDARY OUTCOMES:
Mortality | 3 months
  90-day mortality
Morbidity | 3 months
  90-day morbidity
Colorectal cancer-specific quality of life (EORTC QLQ - CR29) at 1 year | 1 year
  The European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire-Colorectal Cancer (EORTC QLQ-CR29) scale will be recorded preoperatively and at 12 months. Surgical procedures will be compared in terms of improvement in EORTC QLQ-CR29 scores.

CONTACTS AND LOCATIONS:
Overall Officials: Osman Civil, MD, Study Director — Medipol University
Locations (2):
- Turkey (Türkiye) (2):
  - Medipol University Bahcelievler Hospital, Istanbul
  - Medipol Mega Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided